CLINICAL TRIAL: NCT07026630
Title: Validating the Efficacy of Activities of Daily Living (ADL)-Focused Virtual Reality (VR) in Upper-Limb Rehabilitation for Acquired Brain Injury (ABI) Individuals: A Pilot Clinical Trial
Brief Title: Activities of Daily Living (ADL) Virtual Reality (VR) for Acquired Brain Injury (ABI) Upper-Limb Rehabilitation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB disapproved the study protocol on 13-Nov-2025
Sponsor: Indiana University (Other)
Collaborators: Indiana University Health (Other)
Responsible Party: Principal Investigator, Hee-Tae Jung, Assistant Professor, Health Informatics, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23118
Record Dates: First submitted 2025-06-05; First posted 2025-06-18 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Upper Limb Rehabilitation; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- ADL-Focused Virtual Reality (Experimental): Participants will receive 24 one-hour rehabilitation sessions with a licensed occupational therapist trained in stroke recovery and with the VR system. Each therapy session will include range of motion and general strengthening activities as well as 20-30 minutes of the intervention (ADL-focused upper-limb virtual reality training). The goal is to complete rehabilitative training in 12 weeks, with each participant training two times per week.
  Interventions: Device: Cooking In the Kitchen

INTERVENTIONS:
Device: Cooking In the Kitchen — The virtual reality (VR) training tool simulates cooking, an activity of daily living (ADL). The layout of VR environments intentionally place ingredients, tools, and the recipe book far away from the user to require gross upper-limb physical movements. Successful step completion requires reaching to obtain ingredients or turn book pages, grabbing to hold or release objects, and chopping, scooping, stirring, and pouring motions to prepare food items. The VR tool includes three versions of varying graphical complexity: Simple, Standard, and Complex.
  Complexity is controlled by stimuli count and detail level. For example, Simple features an empty room with monotone colors, basic shapes, and no extra features. In contrast, Complex resembles a fully-fledged kitchen with color patterns, textures, background details, and sounds.

SUMMARY:
Acquired brain injury (ABI) individuals have shown greater engagement and functional recovery when trained in virtual reality (VR)-assisted rehabilitation therapies.

After developing an activities of daily living (ADL)-focused VR system in a prior study, this related follow-up study aims to test the efficacy and impact of this VR system on upper-limb rehabilitation outcomes of ABI individuals when routinely integrated into treatment plans.

DETAILED DESCRIPTION:
After completion of informed consent, patients will undergo screening assessments to determine eligibility for study participation.

All eligible participants integrate VR into rehabilitation treatment plans twice per week for 12 weeks. Graphical complexity increases progressively throughout the study: "Simple" in Weeks 1-4, "Standard" in Weeks 5-8, and "Complex" in Weeks 9-12. Assessments are conducted at pre-intervention and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* acquired brain injury with upper extremity impairment
* Fugl-Meyer Assessment of Upper Extremity (FMA-UE) score of 20 points or more
* able to follow commands and instructions
* least 2 months post-stroke, in the subacute or chronic recovery phase

Exclusion Criteria:

- contraindications that increase susceptibility to VR-related adverse events and/or prevent completion of training tasks, such as seizures, epilepsy, visual acuity deficits (besides glasses), vertigo, nystagmus, motion sensitivity, or other non-ABI conditions that impede upper limb movement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment for Upper Extremity | Baseline (pre-intervention), Week 6, and End-of-Study (post-intervention, Week 13)
  The Fugl-Meyer Assessment (FMA) is a physical performance impairment index that evaluates motor recovery.
  Domains of motor function, sensation, balance, range of motion, and pain are measured on a 3-point ordinal scale.
  The upper extremity (UE) section score ranges from 0 to 66, with higher scores indicating less impairment.

SECONDARY OUTCOMES:
Stroke Impact Scale | Baseline (pre-intervention) and End-of-Study (post-intervention, Week 13)
  The Stroke Impact Scale (SIS) holistically evaluates quality of life after a stroke. The SIS-16 version is a self-report questionnaire that assesses the ability to perform daily physical activities on a 5-point Likert scale.
  Score ranges from 0 to 100, with higher scores indicating better capacity and milder stroke impact.
Lawton Instrumental Activities of Daily Living | Baseline (pre-intervention) and End-of-Study (post-intervention, Week 13)
  The Lawton Instrumental Activities of Daily Living (IADL) Scale uses self-reported information to assess performance during independent living. Topics vary and include tasks such as phone use, shopping, housekeeping, and medication management.
  Score ranges from 0 (low function and dependent) to 8 (high function and independent).
  Scoring differs by gender due to known differences in IADL performance.

OTHER OUTCOMES:
Mini-Mental State Examination | Baseline (pre-intervention)
  The Mini-Mental State Examination (MMSE) is an 11-question cognitive performance assessment that evaluates orientation, understanding, language, attention, and memory.

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Tae Jung, Ph.D., Principal Investigator — Indiana University, Luddy School of Informatics, Computing, and Engineering; Peter Altenburger, Ph.D., PT, Principal Investigator — Indiana University, School of Health & Human Sciences; Indiana University Health, Center for Advanced Neurorehabilitation
Locations (1):
- Indiana University Health, Neurorehabilitation & Robotics, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided